CLINICAL TRIAL: NCT05438836
Title: ROAR-A: Re-optimization Based Online Adaptive Radiotherapy of Anal Cancer
Brief Title: Re-optimization Based Online Adaptive Radiotherapy of Anal Cancer
Acronym: ROAR-A
Status: Recruiting | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Eva Serup-Hansen, Clinical oncologist, MD, PhD, Herlev Hospital
Other Study IDs: H-21028093
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Anal Cancer; Anal Carcinoma; Anal Squamous Cell Carcinoma
Keywords: adaptive radiotherapy; Anal cancer; Online Adaptive radiotherapy (oART)
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Online adaptive radiotherapy: Daily online adaptive radiotherapy
  Interventions: Radiation: online adaptive radiotherapy

INTERVENTIONS:
Radiation: online adaptive radiotherapy — Online adaptive radiotherapy compared to standard non-adaptive Image-Guided Radiotherapy
  Other Names: Varian Ethos Adaptive Radiation Therapy

SUMMARY:
A single-arm, prospective, Phase II, single-center clinical trial that will investigate if daily online adaptive radiotherapy for anal cancer will significantly reduce early treatment-related GI toxicity compared with the historically reported rate for non-adaptive intensity modulated radiation therapy (IMRT).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-verified anal cancer
* Eligible for curative intended radiotherapy
* Written and oral consent

Exclusion Criteria:

* Other malignant disease within the past 5 years (excluding basal cell carcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-metastatic squamous cell carcinoma of the anus, referred for chemo-radiotherapy with curative intent.
Sampling Method: Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Early Rate of Common Terminology Criteria for Adverse Events (CTCAE) Gastrointestinal Toxicity grade 2 or more (scale from 0-5, 5 being the highest) | from mid-treatment to 3 months after end of treatment
  percentage of patients with grade 2 or more early treatment-related Gastrointestinal-toxicity

SECONDARY OUTCOMES:
All Early Common Terminology Criteria for Adverse Events (CTCAE) Treatment Related Toxicities. Grade 1-5 (5 being the highest) | from mid-treatment to 3 months after end of treatment
  percentage of patients with grade 2 or more early treatment-related toxicity
All Late Common Terminology Criteria for Adverse Events (CTCAE) Treatment Related Toxicities | From 3 months after end of treatment to 5 years follow-up
  percentage of patients with grade 2 or more late treatment-related toxicity
Patient Reported Outcomes (PRO) | from baseline to 5 years follow-up
  Collection of National Cancer Institute Patient Reported Outcome-Common Terminology Criteria for Adverse Events (NCI PRO-CTCAE) questionnaire (scale from none to a lot) and comparison to Common Terminology Criteria for Adverse Events (CTCAE) and dosimetry data
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Assessment | from baseline to 5 years follow-up
  Collection ofEuropean Organisation for Research and Treatment of Cancer (EORTC) Quality of life questionnaire C30
Progression Free Survival | From time of inclusion to disease progression, assessed up to 5 years follow-up
  Progression free survival (from time of inclusion to disease progression)
Overall Survival | From time of inclusion to death from any cause, assessed up to 5 years follow-up
  Overall survival
Disease Free Survival | From time of inclusion to death from bladder cancer, assessed up to 5 years follow-up
  Disease Free Survival
Treatment Related Hospitalization | From of start of radiation therapy through 5 year follow-up
  Hospitalization due to radiation therapy treatment related toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Eva S Serup-Hansen, MD, PhD, Principal Investigator — Herlev og Gentofte Hospital
Locations (1):
- Oncology dept, Herlev and Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Storm KS, Astrom LM, Sibolt P, Behrens CP, Persson GF, Serup-Hansen E. ROAR-A: re-optimization based Online Adaptive Radiotherapy of anal cancer, a prospective phase II trial protocol. BMC Cancer. 2024 Mar 25;24(1):374. doi: 10.1186/s12885-024-12111-1. PMID 38528456